CLINICAL TRIAL: NCT06694636
Title: Intravascular Radiofrequency Ablation of Sympathetic Nerves for the Treatment of Hepatocellular Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Director of Interventional and Vascular Surgery Department, Zhongda Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024ZDSYLL167-P01
Record Dates: First submitted 2024-07-24; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Sympathetic Nerves; Intravascular Radiofrequency Ablation
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: Enrolled patients will receive intravascular Radiofrequency Ablation of Sympathetic Nerves for the Treatment of Hepatocellular Carcinoma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intravascular Radiofrequency Ablation of Sympathetic Nerves Group (Experimental): Enrolled patients will receive Intravascular Radiofrequency Ablation of Sympathetic Nerves for the Treatment of Hepatocellular Carcinoma
  Interventions: Procedure: endovascular radiofrequency ablation and desympathetic nerve surgery

INTERVENTIONS:
Procedure: endovascular radiofrequency ablation and desympathetic nerve surgery — endovascular radiofrequency ablation and desympathetic nerve surgery

SUMMARY:
Patients who met the inclusion criteria were treated with endovascular radiofrequency ablation and desympathetic nerve surgery. After enrollment, endovascular radiofrequency ablation and desympathetic surgery were performed. After radiofrequency ablation, the safety and efficacy of follow-up treatment will be carried out every 1 month or so, including blood routine, liver and kidney function, tumor indicators, abdominal CT/magnetic resonance, etc.

ELIGIBILITY:
Inclusion Criteria:

* Clinically or pathologically confirmed hepatocellular carcinoma (HCC)
* Locally progressed or distant metastatic unresectable advanced HCC
* Progressed after second-line therapy
* Agree to participate in the study and sign the informed consent form

Exclusion Criteria:

* Not suitable for ablation surgery
* Pregnant, lactating and planning to become pregnant
* Orthostatic hypotension
* Mixed liver cancer
* Intestinal obstruction
* Obvious bleeding tendencies and hematologic diseases
* Acute or severe systemic infection;
* Stroke or transient ischemic attack (TIA) within two weeks;
* Acute coronary syndrome within two weeks;
* Evaluated to be not suitable for this trial by investigators

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
ORR | every month, up to 1 year
  Objective Response Rate

SECONDARY OUTCOMES:
PFS | every month, up to 1 year
  Progression Free Survival
DCR | every month, up to 1 year
  disease control rate

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Gao-Jun, Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided